CLINICAL TRIAL: NCT01928966
Title: Effect of Pumpkin Seeds on the Dietary Fatty Acid Intake and Blood Pressure in Women
Acronym: PSS1
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Advisor left the university and student moved to a clinical track
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: TWU-1PS
Record Dates: First submitted 2013-08-21; First posted 2013-08-27 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Cardiovascular Disease; Blood Pressure
Keywords: dietary fat; fat intake; blood pressure; women; phytoestrogen; pumpkin seeds; cardiovascular disease; heart disease; secoisolariciresinol; monounsaturated fat; polyunsaturated fat; feeding study
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I - Pumpkin Seeds (Active Comparator): First four weeks of study: consume perceived normal diet; Second four weeks of study: receive 1.5 ounces of pumpkin seeds per day for consumption; Third four weeks of the study: consume their perceived normal diet.
  Interventions: Other: Pumpkin Seeds
- Group II - Pumpkin Seeds (Active Comparator): First four weeks of study: consume perceived normal diet; Second four week period: consume perceived normal diet; Third four week period: receive 1.5 ounces of pumpkin seeds per day for consumption.
  Interventions: Other: Pumpkin Seeds

INTERVENTIONS:
Other: Pumpkin Seeds — Participants will be asked to consume 1.5 ounces of raw, unsalted pumpkin seeds per day. The 1.5 ounces will be split in to two servings (each 0.75 ounces).

SUMMARY:
The purpose of this study is to determine if the inclusion of 1.5 ounces of pumpkin seeds per day in the diet of women will alter dietary fatty acid intake or blood pressure.

DETAILED DESCRIPTION:
Cardiovascular disease is the number one cause of morbidity and mortality in United States. Diets high in polyunsaturated and monounsaturated fatty acids have been shown to decrease the risk of cardiovascular disease. Pumpkin seeds are a good source of monounsaturated and polyunsaturated fatty acids. Oil extracted from pumpkin seeds has been shown to lower blood pressure. One purpose of this study is to determine whether eating 1.5 ounces of pumpkin seeds per day will improve polyunsaturated and monounsaturated fatty acid intake in the diet in healthy adult women. Another purpose of this study is to determine whether eating 1.5 ounces of pumpkin seeds a day will lower blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Over the age of 18
* Able to read, write, and speak English
* Able to keep a three-day diet diary
* Willing and able to consume pumpkin seeds

Exclusion Criteria:

* Pregnant or planning to become pregnant
* Allergic to pumpkin seeds
* High blood pressure
* Regularly consuming pumpkin seeds (more than 4 times per month)
* Taking blood pressure medication
* Liver disease
* Kidney disease
* Gastrointestinal disease
* History of bariatric surgery
* History of a major cardiovascular event
* Heart disease
* Currently undergoing cancer treatment (except nonmelanoma cancer)
* Following a weight control diet
* Following a disease specific diet
* Following a vegan diet
* Have a diagnosed eating disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Dietary fatty acid intake | 12 weeks
  The dietary fatty acid intake, specifically monounsaturated and polyunsaturated fatty acids, will be measured three times over the course of a twelve week period to determine if fatty acid intake changed during the intervention.
Blood pressure | 12 weeks
  Blood pressure will be measured at every meeting to determine if the addition of pumpkin seeds to the diet altered blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: John D Radcliffe, PhD, Study Chair — Texas Woman's University
Locations (1):
- Texas Woman's University, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The study was stopped before data collection began - no data to share.